CLINICAL TRIAL: NCT00862758
Title: Emergency IND for Provision of Tocilizumab
Brief Title: Request for Single Patient IND for Compassionate/Emergency Use of Tocilizumab
Status: No longer available | Type: Expanded Access
Sponsor: University of Oklahoma (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: 14524
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: juvenile idiopathic arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — 8 mg/kg would be administered IV every 2 weeks for six weeks.

SUMMARY:
Application for Compassionate Use of Tocilizumab in a Boy with Severe Polyarticular Juvenile Idiopathic Arthritis (JIA) Unresponsive to All Licensed Medications.

DETAILED DESCRIPTION:
This trial is for a single subject with juvenile idiopathic arthritis unresponsive to all licensed treatments for JIA, and some licensed only for rheumatoid arthritis. He is currently wheelchair bound and completely dependent for activities of daily living and self-care. He is in constant pain, has abundant warmth and swelling of nearly all joints including TMJs, neck, shoulders, elbows, wrists, MCP and finger joints (even some DIP joints), hips, knees, ankles, subtalar and intertarsal joints, MTP and IP joints of the toes.

Drug at a dose of 8 mg/kg would be administered IV every 2 weeks, with close safety and monitoring studies.

Treatment would be monitored every 2 weeks. Efficacy will be measured using the ACR Pedi 30, 50 and 90 definitions as previously published, based on: 1) physician global assessment of disease activity; 2) parent/patient assessment of overall well-being; 3) functional ability; 4) number of joints with active arthritis; 5) number of joints with limited range of motion; and 6) erythrocyte sedimentation rate.

ELIGIBILITY:
Inclusion Criteria:

* Subject X, polyarticular JIA, not responding to any other drug

Exclusion Criteria:

* Not identified subject

Ages: 11 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen O'Neil, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States